CLINICAL TRIAL: NCT03870204
Title: Validation of the Schistosomiasis Point-of-Care Circulating Cathodic Antigen (POC-CCA) Rapid Urine Test for Qualitative Detection of Schistosoma Japonicum
Brief Title: Validation of POC-CCA Rapid Urine Test for Qualitative Detection of Schistosoma Japonicum
Acronym: SchisCCA
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: INA105; U1111-1263-2399 (Other: WHO UTN Number)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Aged ≥2 Years in Schistosomiasis Affected Areas
Keywords: Schistosoma japonicum
MeSH Terms: conditions — Schistosomiasis japonica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and stool at visit 1 and 3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: POC-CCA rapid urine test — Fresh urine samples will be tested by POC-CCA
  Other Names: Kato-Katz, ELISA, and PCR

SUMMARY:
This is a longitudinal cohort study that will be coordinated with the 2019 schistosomiasis stool survey in Napu. The study will use the stool survey results as entry criteria to identify subjects to become the index cases. Contact investigation will be conducted to the index cases during home visit (Visit 1). The index cases and their contacts meeting the study's eligibility criteria will be recruited. For Visit 1, they will be tested for schistosomiasis by on the spot POC-CCA, stool samples will be tested for KK at Donggala R&D Center Laboratory and urinary tract infection (UTI) by urine dipsticks, stool samples will be tested for schistosomiasis and soil transmitted helminths (STH) by KK at Donggala R&D Center Laboratory and by molecular assay (Taqman qPCR) at the INA-RESPOND Reference Laboratory, while dried blood spots samples will be tested for schistosome antibodies by ELISA at the INA-RESPOND Reference Laboratory. The study KK and/or POC-CCA will be used to determine their schistosomiasis status. Those with positive schistosomiasis status by KK and/or POC-CCA will continue follow up to Visit 2 and 3.

DETAILED DESCRIPTION:
Indonesia's plan for elimination of schistosomiasis by 2025 requires a better understanding of the factors associated with infection, effective epidemiologic monitoring, and optimization of diagnostic and treatment strategies. In settings of low prevalence such as Lindu, Napu and Bada regions of Central Sulawesi, an ultrasensitive technique to diagnose Schistosoma japonicum is needed. A diagnostic test that is efficient, accurate and easy to use would facilitate collection of reliable epidemiologic information and provide and effective means of assessing the impact of mass drug administration (MDA).

Primary Objective:

To estimate the accuracy of the schistosomiasis point-of-care circulating cathodic antigen (POC CCA) urine test for monitoring S. japonicum infection.

Secondary Objective

1. To assess rates of positive testing by POC-CCA rapid urine test, serology, and molecular methods (PCR).
2. To evaluate the impact of abnormal urinary findings, i.e. hematuria and markers of urinary tract infections (UTI), to POC-CCA rapid urine test results.
3. To evaluate the efficacy of praziquantel administered by local primary health centers (Puskesmas).
4. To assess number of schistosome infection using serology and molecular (PCR) as additional tests to disambiguate discordant results between KK and POC-CCA.
5. To assess risk factors related to human schistosome infections.
6. To estimate the proportion of soil transmitted helminths infection (STH), i.e. roundworms (Ascaris lumbricoides), whipworms (Trichuris trichiura), and hookworms (Necator americanus and Ancylostoma duodenale) in this population.
7. To assess the association between color intensity of the POC-CCA rapid urine test band and the schistosome eggs per gram (EPG) of stool.
8. To assess antibody response to schistosome infection. The number in the positive KK group will be 40 subjects, with the lowest estimated number is 25 subjects. Additional positive KK based on the re-testing KK results are expected and should increase the size for the positives. For the negatives, we calculated that a ratio of 4:1 negative to positive will be the best fit, thus 160 negative KK subjects will be enrolled. Additional 20% buffer to the negatives (32 negative KK subjects) will also be needed to estimate the specificity of POC-CCA with acceptable 95% CI. In total, we will enroll between 217 to 232 subjects in this study. The study will enroll all positive cases detected by the 2019 stool survey in Napu until the minimum sample size needed is met or until the data collection period has ended.

ELIGIBILITY:
Inclusion Criteria:

* Reside in schistosomiasis affected areas for at least 8 weeks.
* Age ≥2 years.
* Provides a documented informed consent for participants' ≥18 years old or informed consent by parents/legally accepted representative (LAR) or assent for minor participants prior to the study procedures.
* Willing to comply with the study procedures.
* Agrees to the collection and storage of specimens.

Exclusion Criteria:

None.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Schistosomiasis affected areas are in Lindu, Napu and Bada Valley of Central Sulawesi, Indonesia.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
To estimate the accuracy of the schistosomiasis point-of-care circulating cathodic antigen (POC CCA) urine test for monitoring Schistosoma japonicum infection | 1 year
  * Sensitivity will be established as the proportion of positives that are correctly identified by the POC-CCA rapid urine test, when compared to the Reference Method.
  * Specificity will be established as the proportion of negatives that are correctly identified by the POC-CCA rapid urine test, when compared to the Reference Method.

SECONDARY OUTCOMES:
To assess rates of positive testing by POC-CCA rapid urine test, serology, and molecular methods (PCR). | 1 year
  Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of the POC-CCA rapid urine test.
To evaluate the impact of abnormal urinary findings, i.e. hematuria and markers of urinary tract infections (UTI), to POC-CCA rapid urine test results. | 1 year
  Sensitivity and specificity of the POC-CCA rapid urine test, when compared to the Reference Method, among individuals with abnormal urinary findings.
To evaluate the efficacy of praziquantel administered by local primary health centers (Puskesmas). | 1 year
  Evaluation of cure rate (percentage negative) after praziquantel administration to positive cases by either POC-CCA rapid urine test and/or KK.
To assess number of schistosome infection using serology and molecular (PCR) as additional tests to disambiguate discordant results between KK and POC-CCA. | 1 year
  Number of schistosome infection using serology and molecular as additional examination to disambiguate discordant findings between KK and POC-CCA.
To assess risk factors related to human schistosome infections. | 1 year
  Risk factors will be determined by estimating the odds ratio for each potential risk factor against the Reference Method results.
To estimate the proportion of soil transmitted helminths infection (STH), i.e. roundworms (Ascaris lumbricoides), whipworms (Trichuris trichiura), and hookworms (Necator americanus and Ancylostoma duodenale) in this population. | 1 year
  Proportion of soil transmitted helminth infections
To assess the association between color intensity of the POC-CCA rapid urine test band and the schistosome eggs per gram (EPG) of stool. | 1 year
  Association between the color intensity of the POC-CCA rapid urine test and the schistosome EPGs of stool.
To assess antibody response to schistosome infection. | 1 year
  Antibody response to schistosome infection.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Karyana, dr. MKes, Principal Investigator — Ina-Respond
Locations (1):
- Donggala Research and Development (R&D) Center, Ministry of Health of Indonesia, Donggala, Central of Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Currently we not have any plan to share IPD.